CLINICAL TRIAL: NCT01640548
Title: A Retrospective Chart Review on the Use of Biologics in Monotherapy for the Treatment of Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28372
Record Dates: First submitted 2012-07-06; First posted 2012-07-13 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional, retrospective, cross sectional chart review study will evaluate the management of rheumatoid arthritis patients with a biologic in monotherapy. Data from eligible patients will be collected from the patient's last visit on the prior rheumatoid arthritis treatment and from the most recent visit for the biological monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of rheumatoid arthritis by a Rheumatologist
* Patient being prescribed with a biologic in monotherapy

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a biologic in monotherapy for rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United Kingdom (26):
  - Abergavenny
  - Basildon
  - Basingstoke
  - Belfast
  - Blackburn
  - Bournemouth
  - Cambridge
  - Cannock
  - Dewsbury
  - Dudley
  - Durham
  - Eastbourne
  - Edinburgh
  - Glasgow
  - Greenock
  - Harlow
  - Inverness
  - Kirkcaldy
  - London
  - Portsmouth
  - Sheffield
  - Truro
  - Warrington
  - Westbury-on-Trym, Bristol
  - Wigan
  - Wolverhampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis (RA) Cohort: Participants on biologic disease modifying anti-rheumatic drug (bDMARD) monotherapy for RA and on any RA treatment in the past were observed and data was collected retrospectively from a chart review for approximately 9 months.
Period: Overall Study
Arm/Group | Rheumatoid Arthritis (RA) Cohort
Started | 309
Completed | 309
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Included all the participants who entered the retrospective chart review.
Groups:
- Rheumatoid Arthritis Cohort: Participants on bDMARD monotherapy for RA and on any RA treatment in the past were observed and data was collected retrospectively from a chart review for approximately 9 months.
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11.99)
Gender [Count of Participants; unit: Participants]
  Female | 224
  Male | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Participants Receiving Biologic Disease Modifying Anti-Rheumatic Drugs (bDMARDs) in Monotherapy as Current Treatment for RA According to National Institute for Health and Clinical Excellence (NICE) Guidelines by Type of bDMARD
Description: bDMARDS for RA treatment include etanercept, adalimumab, tocilizumab, rituximab, certolizumab pegol, infliximab, golimumab, abatacept and anakinra medications. Current bDMARDs were defined as those with a start date on or after the date of collection, or those with a start date before the date of collection and an end date on or after the date of collection. NICE guidelines recommend the participants with severe active RA who inadequately responded to prior DMARD treatment (trial of 2 DMARDs, one which includes methotrexate) and were intolerant to methotrexate or the treatment with methotrexate considered inappropriate be treated with a biologic DMARD monotherapy.
Time Frame: 9 months
Population: Included all the participants who entered the retrospective chart review.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 309
percentage of participants
  Etanercept | 39.5
  Adalimumab | 28.8
  Tocilizumab | 12.3
  Rituximab | 10.7
  Certolizumab Pegol | 6.1
  Infliximab | 1.0
  Golimumab | 1.0
  Abatacept | 0.6

2. Primary Outcome: Percentage of Participants Treated With Traditional DMARDs as Their Previous Treatment for RA by Type of DMARD
Description: Traditional DMARDS for RA treatment include methotrexate, sulfasalazine, leflunomide, hydroxychloroquine, gold compounds, penicillamine, cyclosporine, azathioprine, chlorambucil, mercaptopurine, and mycophenolate mofetil medications. Previous RA treatment included all the treatments received prior to switching to current RA treatment.
Time Frame: 9 months
Population: Included all the participants who took any past traditional DMARDs.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 303
percentage of participants
  Methotrexate | 94.7
  Sulfasalazine | 78.9
  Leflunomide | 46.9
  Hydroxychloroquine | 42.9
  Gold Compounds | 29.4
  Penicillamine | 9.9
  Cyclosporine | 9.2
  Azathioprine | 8.9
  Chlorambucil | 0.3
  Mercaptopurine | 0.3
  Mycophenolate Mofetil | 0.3

3. Primary Outcome: Percentage of Participants With bDMARD and Concomitant Traditional DMARD Regimen as Previous RA Treatment at Anytime Prior to Switch to bDMARD Monotherapy by Type of bDMARD
Description: bDMARDS for RA treatment include etanercept, adalimumab, tocilizumab, rituximab, certolizumab pegol, infliximab, golimumab, abatacept and anakinra medications. Only the most frequently used (> 10% of participants) bDMARDs with concomitant traditional DMARD as previous treatment for RA were reported. If a participant was recorded to have been treated with a single bDMARD more than once, the participant was counted only once per type of bDMARD. If participant received 2 different types of bDMARDs as part of their previous treatment, the participant was counted twice, once per each type of bDMARD; therefore, the percentage of participants did not add up to 100%.
Time Frame: 9 months
Population: Included participants who were previously treated with any bDMARD with concomitant traditional DMARD prior to switch to bDMARD monotherapy as current RA treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 131
percentage of participants
  Etanercept | 51.9
  Adalimumab | 45.0
  Rituximab | 16.8
  Infliximab | 15.3
  Tocilizumab | 9.2
  Abatacept | 1.5
  Anakinra | 0.8

4. Primary Outcome: Percentage of Participants With bDMARD Monotherapy as Previous RA Treatment at Anytime Prior to Switch to bDMARD Monotherapy
Description: bDMARDS for RA treatment include etanercept, adalimumab, tocilizumab, rituximab, certolizumab pegol, infliximab, golimumab, abatacept and anakinra medications. Only the most frequently used (> 10% of participants) bDMARDs in monotherapy as previous treatment for RA were reported. If a participant was recorded to have been treated with a single bDMARD more than once, the participant was counted only once per type of bDMARD. If participant received 2 different types of bDMARDs as part of their previous treatment, the participant was counted twice, once per each type of bDMARD; therefore, the percentage of participants did not add up to 100%.
Time Frame: 9 months
Population: Included participants who received bDMARD as monotherapy as previous treatment prior to switch to bDMARD monotherapy as current treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 117
percentage of participants
  Etanercept | 53.0
  Adalimumab | 41.9
  Certolizumab Pegol | 13.7
  Rituximab | 11.1
  Tocilizumab | 6.0

5. Secondary Outcome: Assessment of Disease Activity Score of 28 Joint Count (DAS28) by Either Erythrocyte Sedimentation Ratio (ESR) or C-Reactive Protein (CRP)
Description: DAS28 was calculated from the tender joint count (TJC) of 28 joints, swollen joint count (SJC) of 28 joints, ESR (in millimeters/hour) or CRP (in milligrams/liter), and the participant's global assessment of disease activity (visual analog scale: 0=no disease activity to 100=maximum disease activity). The formula for calculating DAS28 score using ESR value is: 0.56 x square root (√) of TJC + 0.28 x √(SJC) + 0.70 x log natural (ESR) + 0.014 x global assessment of RA score. The formula for calculating DAS28 score using CRP value is: 0.56 x √(TJC) + 0.28 x √(SJC) + 0.36 x log natural (CRP+1) + 0.014 x global assessment of RA score +0.96. The DAS28 score range was 0-9.4 where higher scores represented higher disease activity.
Time Frame: 9 months
Population: Included the number of participants who were evaluable for DAS28 assessment. "n" represents the number of participants who were evaluable for that particular assessment.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 149
scores on a scale
  ESR-DAS28 score (n=149) | 3.41 [3.16 to 3.66]
  CRP-DAS28 score (n=72) | 3.21 [2.84 to 3.58]

6. Primary Outcome: Percentage of Participants With Concomitant Treatment Other Than DMARDs for RA by Type of Treatment
Description: All corticosteroids and non-steroidal anti-inflammatory drugs taken as previous and current treatments for RA were coded according to the Roche international non-proprietary name dictionary.
Time Frame: 9 months
Population: Included all the participants who entered the retrospective chart review.
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 309
percentage of participants
  Participants with any previous treatment for RA | 96.1
  Non-steroidal anti-inflammatories | 83.8
  Corticosteroids | 77.3

7. Secondary Outcome: Total Number of Tender Joints and Swollen Joints and Non-Evaluable DAS 28 Joints When Assessed Using Both ESR and CRP Methods
Description: DAS28 was calculated from the tender joint count (TJC) of 28 joints, swollen joint count (SJC) of 28 joints, ESR (in millimeters/hour) or CRP (in milligrams/liter), and the participant's global assessment of disease activity (visual analog scale: 0=no disease activity to 100=maximum disease activity). TJC and SJC assessed as part of the DAS28 outcome measure assessment were reported.
Time Frame: 9 months
Population: Includes all participants who were evaluable for this outcome. "n" represents the number of participants who were evaluable for that particular assessment.
Measure: Mean (95% Confidence Interval); unit: joints count
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 164
joints count
  ESR-TJC (n=164) | 3.2 [2.4 to 4.0]
  ESR-SJC (n=163) | 1.6 [1.2 to 2.0]
  ESR-Non-evaluable DAS28 joints (n=125) | 0.4 [0.1 to 0.8]
  CRP-TJC (n=73) | 3.7 [2.4 to 4.9]
  CRP-SJC (n=74) | 2.3 [1.5 to 3.2]
  CRP-Non-evaluable DAS28 joints (n=30) | 0.5 [0.2 to 0.8]

8. Primary Outcome: Percentage of Participants by Reason for Choosing Previous and Current bDMARDs in Monotherapy
Description: Both previous and current bDMARDs were presented together for each subgroup, therefore the percentage of participants under each reason did not add up to 100%.
Time Frame: 9 months
Population: Included all participants who entered the retrospective chart review.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 309
percentage of participants
  Physician's preference/experience/Unknown | 84.1 [79.6 to 88.0]
  Participant preference | 5.8 [3.5 to 9.1]
  Contra-indication to alternative drug | 4.9 [2.7 to 7.9]
  Other | 8.4 [5.6 to 12.1]

9. Secondary Outcome: Duration of Treatment With the Current bDMARD Usage in Monotherapy
Time Frame: 9 months
Population: Included all participants who received bDMARD monotherapy as their current treatment for RA. "n is the number of participants who received that particular bDMARD as their current RA treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 308
months
  Abatacept (n=2) | 38.70 [10.3 to 67.1]
  Adalimumab (n=89) | 41.70 [1.1 to 148.2]
  Certolizumab Pegol (n=19) | 13.20 [1.1 to 26.0]
  Etanercept (n=121) | 36.20 [1.7 to 145.1]
  Golimumab (n=3) | 6.60 [0.8 to 20.3]
  Infliximab (n=3) | 13.60 [0.2 to 32.0]
  Rituximab (n=33) | 18.20 [1.1 to 71.1]
  Tocilizumab (n=38) | 12.05 [0.1 to 54.7]

10. Secondary Outcome: Duration of Treatment With bDMARDs in Monotherapy as Previous Treatment for RA
Time Frame: 9 months
Population: Included participants treated with a bDMARD monotherapy as previous treatment for RA prior to switch to current bDMARD monotherapy. "n" is the number of participants who received particular bDMARD as previous RA treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 117
months
  Adalimumab (n=56) | 8.55 [0.4 to 102.5]
  Certolizumab Pegol (n=16) | 0.90 [0.6 to 12.0]
  Etanercept (n=82) | 10.50 [0.5 to 123.0]
  Rituximab (n=14) | 4.25 [0.5 to 44.0]
  Tocilizumab (n=7) | 7.80 [0.9 to 14.1]

11. Secondary Outcome: Duration of Treatment of bDMARD Administered With Concomitant Traditional DMARD as Previous Treatment for RA
Time Frame: 9 months
Population: Included participants who were treated with a bDMARD with concomitant traditional DMARD as previous treatment for RA. "n" is the number of participants who received particular bDMARD as previous RA treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Rheumatoid Arthritis Cohort
Number analyzed (Participants) | 131
months
  Abatacept (n=2) | 4.10 [2.9 to 5.3]
  Adalimumab (n=62) | 18.60 [1.2 to 107.9]
  Anakinra (n=1) | 9.50 [9.5 to 9.5]
  Etanercept (n=72) | 15.95 [0.7 to 87.2]
  Infliximab (n=21) | 10.00 [0.0 to 106.3]
  Rituximab (n=41) | 0.00 [0.0 to 37.2]
  Tocilizumab (n=15) | 3.40 [0.0 to 31.6]

ADVERSE EVENTS:
Time Frame: 9 months
Description: Adverse events data were collected retrospectively for participants treated with rituximab or tocilizumab only.
Arm/Group | Rheumatoid Arthritis Cohort
Serious Adverse Events (participants affected / at risk) | 3/71
Other Adverse Events (participants affected / at risk) | 6/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Cohort (N=71)
Lower Respiratory Tract Infection (Infections and infestations) | 1
Necrotising fascitis (Infections and infestations) | 1
Cholecystitis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis Cohort (N=71)
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.